CLINICAL TRIAL: NCT03688269
Title: Determination of the Minimal Effective Concentration (EC90) of Ropivacaine in Axillary Brachial Plexus Block With Intravenous Dexamethasone or Saline Injection
Brief Title: Minimal Effective Concentration (EC90) of Ropivacaine
Acronym: AxiRopiDexa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P/2018/384
Record Dates: First submitted 2018-09-14; First posted 2018-09-28 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia, Conduction; Ropivacaine; Dexamethasone; Axillary Brachial Plexus Block
Keywords: regional anesthesia; dexamethasone; ropivacaine

STUDY DESIGN:
Intervention Model Description: allocation to one of the 2 arm after randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous dexamethasone (Experimental): Axillary Brachial Plexus Block with perineural Ropivacaine. Concentration determined by sequential up and down method.
  Intravenous injection of 8mg/2ml Dexamethasone during the regional anesthesia
  Interventions: Drug: Intravenous dexamethasone; Drug: Perineural ropivacaine
- Intravenous saline (Placebo Comparator): Axillary Brachial Plexus Block with perineural Ropivacaine. Concentration determined by sequential up and down method.
  Intravenous injection of 2ml Saline 0.9% during the regional anesthesia
  Interventions: Drug: Intravenous saline; Drug: Perineural ropivacaine

INTERVENTIONS:
Drug: Intravenous dexamethasone — Intravenous injection of 8mg/2ml dexamethasone
  Arms: Intravenous dexamethasone
Drug: Intravenous saline — Intravenous injection of 2ml Saline 0.9%
  Arms: Intravenous saline
Drug: Perineural ropivacaine — Perineural injection of 20ml ropivacaine with adjustment of the concentration determined by sequential up and down method

SUMMARY:
Prospective up and down sequential evaluation of the minimal effective concentration of perineural ropivacaine for 90% success in axillary brachial plexus block with the injection of intravenous dexamethasone or saline placebo during regional anesthesia performance

DETAILED DESCRIPTION:
ropivacaine concentration determined by up and down sequential method dexamethasone or saline placebo determined by randomisation

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* ASA Score 1,2 et 3 (American Society of Anesthesiologists Score)
* surgery under axillary brachial plexus block
* signed information consent

Exclusion Criteria:

* pregnancy and breastfeeding
* contraindication to regional anesthesia or technical impossibility
* impaired coagulation
* delay of surgery to short to allow regional anesthesia
* dementia or under administrative supervision
* allergy and contraindication to dexamethasone or ropivacaine
* total dose of ropivacaine higher than 3 mg / kg (recommended dose for upper limb regional anesthesia)
* opioids or pain killers abuse or addiction
* steroids consumption in the past 6 months
* surgery estimated to be greater than 4 hours
* anticipated bad observation of treatment
* patient enrolled in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Surgical Effectiveness of regional anesthesia at 30min | Time of surgery
  Ability to perform surgery under regional anaesthesia without supplementary anaesthesia

SECONDARY OUTCOMES:
time between regional anesthesia and surgical incision | Time of surgery
  time between the end of regional anesthesia and the beginning of surgical incision
Effectiveness of regional anaesthesia on Pin-Prick sense | Time of anaesthesia
  Defined by a loss of pain sensation at the pinprick test at 30min after the end of regional anaesthesia
Effectiveness of regional anaesthesia on cold sensation | Time of anaesthesia
  Defined by a loss of sensation of cold application on skin at 30min after the end of regional anaesthesia
Effectiveness of regional anaesthesia on motor function | Time of anaesthesia
  Defined by a paresis at 30min after the end of regional anaesthesia (modified bromage score)
recovery of regional anesthesia: pain | first 48h
  time to first pain sensation in the surgical wound after the end of regional anaesthesia
recovery of regional anesthesia: motor | first 48h
  time to motor recovery of the arm after the end of regional anaesthesia
recovery of regional anesthesia: sensory | first 48h
  time to sensory recovery of the arm after the end of regional anaesthesia
complication related to regional anesthesia and/or intravenous dexamethasone | month 6
  any complication during the first 6 month after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Francis BERTHIER, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing in progress in the institution